CLINICAL TRIAL: NCT03202069
Title: Effect of Daily Protein Intake Patterns During Weight Loss on Dietary Adherence and Body Composition in Women
Brief Title: Protein Eating Patterns and Weight Loss
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: USDA Grand Forks Human Nutrition Research Center (U.S. Federal Agency)
Collaborators: North Dakota Beef Commission (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: GFHNRC510
Record Dates: First submitted 2017-06-26; First posted 2017-06-28 (Actual); Last update posted 2025-04-16 (Actual); Status verified 2025-04

CONDITIONS: Obesity
Keywords: Protein; Weight Loss
MeSH Terms: conditions — Obesity; Weight Loss

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Even protein intake (Experimental): Menu to provide 90 g of protein per day in an even distribution of 30 g at each meal.
  Interventions: Other: Even protein
- Skewed protein intake (Experimental): Menu to provide 90 g of protein per day in a skewed distribution of 10 g at breakfast, 15 g at lunch and 65 g at dinner.
  Interventions: Other: Skewed protein

INTERVENTIONS:
Other: Even protein — Intake of even protein 5 day rotating menu
  Arms: Even protein intake
Other: Skewed protein — Intake of skewed protein 5 day rotating menu
  Arms: Skewed protein intake

SUMMARY:
The purpose of this study is to determine the effects of daily protein intake patterns on body composition and eating behaviors during weight loss.

DETAILED DESCRIPTION:
The reinforcing value of food varies greatly among individuals, but is strongest for those who are overweight or obese. Reducing energy intake, which is necessary for overweight and obese individuals to achieve a healthier body weight, increases the reinforcing value of food - especially for energy-dense snack foods. Food is a powerful reinforcer and is associated with energy intake; making it a primary contributing factor to an individual's weight loss struggle. Developing a way to decrease or limit the increase in food reinforcement during energy deficits would have important clinical impact. High-protein diets are known to be efficacious for weight loss and recently have been shown to decrease stimulation of the reward areas of the brain that stimulate reward-driven eating behavior. Nonetheless, sustaining a high-protein diet can be difficult, especially for women. Consuming a modest amount of protein at each meal may be better tolerated. However, we do not know whether this pattern of protein intake can assist women in staying "on track" with weight loss goals. This study will help begin to elucidate the connections between the daily pattern of protein intake on diet adherence, alterations in food reinforcement, and favorable body composition changes during weight loss.

ELIGIBILITY:
Inclusion Criteria:

* BMI 28-45 kg/m2

Exclusion Criteria:

* unable or unwilling to consume animal products
* unable or unwilling to attend treatment group meetings
* had more than a 10% change in body weight in the 2 months prior to study start date
* consuming a specialized diet
* have a history of and eating or gastrointestinal disorder
* currently or planning on becoming pregnant during the study timeline
* lactating
* have an uncontrolled metabolic illness/disease (fasting glucose >125 mg/dL)
* have uncontrolled hypertension (>160/99 mm Hg)
* have cancer or in short-term remission (less than 3 years)
* have an infectious disease
* suffer from alcohol or drug abuse
* use tobacco and/or e-cigarette products on a regular basis
* taking medications known to affect energy expenditure and appetite

Ages: 20 Years to 44 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 45 (Actual)
Dates: Start 2017-10-02 (Actual); Primary Completion 2023-04-14 (Actual); Study Completion 2023-04-14 (Actual)

PRIMARY OUTCOMES:
Body Composition | 8 and 16 weeks
  Determine the effects of two patterns of daily protein intake on changes in fat mass and fat-free mass during weight loss.
Diet Adherence | 16 weeks
  Determine the effects of two patterns of daily protein intake on weight loss diet adherence and putative mediators (satisfaction, satiety, hunger, and reinforcing value of energy dense foods) of adherence.

SECONDARY OUTCOMES:
Barriers to weight control | 1 hour
  Nominal Group Technique results providing an exhaustive list of barriers to weight control in overweight and obese women
Change in skeletal muscle protein breakdown | 8 and 16 weeks
  The effect of consuming two patterns of daily protein intake on 3-Methylhistidine degradation, a biochemcial marker of skeletal muscle protein breakdown
Circulating carotenoid levels | 8 and 16 weeks
  The effect of consuming two patterns of protein intake during weight loss on circulating carotenoid levels.
Relative reinforcing value (RRV) of food | 8 and 16 weeks
  The effect of consuming two patterns of daily protein intake during weight loss on the RRV of energy-dense snack food
Change in bone turnover | 8 and 16 weeks
  The effect of consuming two patterns of daily protein intake during weight loss on osteocalcin, alkaline phosphatase, acid phosphatase, and collagen cross-link molecules -- biochemical markers of bone formation and resorption
Plasma lipids | 8 and 16 weeks
  The effect of consuming two patterns of daily protein intake during weight loss on lipid and triglyceride molecular speciation.

CONTACTS AND LOCATIONS:
Overall Officials: Shanon Casperson, PhD, Principal Investigator — USDA Grand Forks Human Nutrition Research Center
Locations (1):
- USDA Grand Forks Human Nutrition Research Center, Grand Forks, North Dakota, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] De Leon A, Roemmich JN, Casperson SL. Daily Dietary Protein Distribution Does Not Influence Changes in Body Composition During Weight Loss in Women of Reproductive Years with Overweight or Obesity: A Randomized Controlled Trial. J Nutr. 2024 Apr;154(4):1347-1355. doi: 10.1016/j.tjnut.2024.02.009. Epub 2024 Feb 15. PMID 38365118
- See also: Grand Forks Human Nutrition Research Center Current Nutrition Studies — https://www.ars.usda.gov/plains-area/gfnd/gfhnrc/docs/nutrition-studies/nutrition-studies/

DOCUMENTS (1):
  • Informed Consent Form (2023-01-27): https://cdn.clinicaltrials.gov/large-docs/69/NCT03202069/ICF_000.pdf